CLINICAL TRIAL: NCT01391234
Title: Phase II Pilot Single Arm Prospective Clinical Trial of Rapid Institution of Helical TomoTherapy-based Radiation Therapy for Patients With Painful Osseous Metastatic Disease
Brief Title: Rapid Radiation Therapy for Painful Osseous Metastatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Paul W. Read, MD, Study Chair, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15625
Record Dates: First submitted 2011-06-14; First posted 2011-07-11 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Bone Metastases
Keywords: Metastatic bone disease; Bone metastases; Radiation therapy; TomoTherapy
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STAT RT planning and delivery workflow (Experimental): single arm
  Interventions: Radiation: STAT RT planning and delivery workflow

INTERVENTIONS:
Radiation: STAT RT planning and delivery workflow — * Patients will receive simulation, planning, quality assurance, and their first treatment in a single day using the STAT RT workflow.
  * Patients will receive a total of 1-5 fractions of high dose palliative radiation therapy via TomoTherapy consisting of 5-10 Gray per fraction.
  * Data will be collected to evaluate the effectiveness of our novel image co-registration techniques, CT-detector-based exit dose calculations, and infrared patient position monitoring. These novel techniques for image co-registration, radiation dose calculations, and patient position monitoring will not alter or replace standard of care techniques.
  Other Names: TomoTherapy-based Radiation Therapy

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of an experimental workflow that may result in a faster way to plan and deliver radiation for the treatment of pain caused by metastatic bone tumors (tumors that originally came from another organ and have spread to bones causing pain) or multiple myeloma (a type of cancer that begins in white blood cells that produce antibodies).

The current standard of care radiation treatment planning and delivery takes 2 to 3 weeks from start to finish. The investigators have developed an experimental workflow: a radiation treatment planning and delivery workflow called "STAT RT" (STAT means "right away", and RT means radiation therapy). This experimental workflow may shorten the time it takes to plan and treat painful bone metastases to 1 week or less. All steps in this process will be performed within the current standard of care but in a shorter time frame to allow treatment to start sooner.

The investigators will evaluate effectiveness by requesting patients to complete pain and quality of life questionnaires before and after treatment. The investigators will also be collecting additional information from their treatments that will help us make future workflows even more efficient.

DETAILED DESCRIPTION:
Background: Osseous metastatic disease causes significant pain, decreased functioning, and decreased quality of life. Progressive bone destruction can lead to pathologic fractures or spinal cord compression leading to orthopedic surgery, paralysis, and/or patients becoming bedridden. Opioids can alleviate pain but have neurologic and gastrointestinal side effects that further decrease quality of life. Radiation therapy can effectively reduce pain and opioid use and prevent further bone destruction, however, its use is limited because the current workflow frequently requires one week for planning and two weeks for delivery. Additionally, typical palliative radiation plans for osseous metastases lack conformality of dose to the tumor volume, and therefore, result in radiation-induced toxicity to large volumes of adjacent normal tissue. Recent software and hardware advancements provide the opportunity to revolutionize the palliative treatment of osseous metastases. The investigators propose to investigate a novel TomoTherapy-based workflow, called STAT RT, which includes same day CT simulation, treatment planning, and quality assurance measurements coupled with highly conformal treatment delivery for patients with osseous metastases in a pilot clinical trial.

Objective: The overall goal of this STAT RT proposal is to develop a more rapid, convenient, and effective palliative radiation approach for patients with osseous metastases that is less toxic and less expensive than current treatment regimens. The investigators have already optimized the conformality of TomoTherapy-based radiation doses for osseous metastases, and the investigators have developed a STAT RT workflow that condenses standard of care simulation, planning, quality assurance, and treatment delivery into 5-6 hours. Additional optimization and integration of new radiation therapy computing processes will allow for real time simulation, planning, and delivery via a novel Scan-Plan-Treat STAT RT workflow that will ultimately require only 30 minutes. In this study the investigators will evaluate the effectiveness of the current STAT RT workflow, and the investigators will investigate techniques for further optimization that will be needed to create a 30 minute Scan-Plan-Treat STAT RT workflow.

Primary Specific Aim/ Hypothesis: The investigators will quantify the time for pain relief, amount of pain relief, opioid use reduction, functional scores, quality of life, and satisfaction of patients treated with STAT RT for osseous metastases. The investigators hypothesize that these patients will have rapid and significant pain relief, improved quality of life, and high patient satisfaction.

Secondary Specific Aim/ Hypothesis: The investigators will optimize the integration of commercially available and in-development software to develop the Scan-Plan-Treat STAT RT workflow. Specifically, the investigators will A) optimize rigid and deformable co-registration of pre-contoured diagnostic image sets to MVCT simulation scans and compare the accuracy to the same pre-contoured diagnostic image sets co-registered to kilovoltage CT (kVCT) simulation images and then kVCT simulation to MVCT scan co-registration, B) optimize CT-detector-based exit dose measurement algorithms for quality assurance and compare to standard of care phantom-based quality assurance, C) optimize the accuracy of an in-house real time infrared tracking system for intrafractional patient position monitoring to ensure accurate patient treatment. The investigators hypothesize that these new components will provide effective and efficient methods for treatment planning, quality assurance, and patient position monitoring that can be used in a future 30 minute Scan-Plan-Treat STAT RT workflow.

Study design: The investigators will recruit 30 cancer patients with 1-3 painful osseous metastatic lesions (target sites) who are candidates for palliative radiation therapy. Patients will receive 1-5 fractions of 5-8 Gray (Gy) (minimum biologic effective dose of 25 Gy) of conformal radiation therapy delivered to the target sites via the Helical TomoTherapy system using the STAT RT workflow. Data will be collected to evaluate the effectiveness of our novel image co-registration techniques, CT-detector-based exit dose calculations, and infrared patient position monitoring. These novel techniques for image co-registration, radiation dose calculations, and patient position monitoring will not alter or replace standard of care techniques. Using validated surveys the investigators will record patient pain, analgesic use, function, quality of life, and patient satisfaction prior to treatment and at 1 week, 4 weeks, 8 weeks, 12 weeks, 6 months, and 12 months after therapy. Radiation-induced treatment related toxicities will be captured during treatment and at the above time points.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a biopsy proven diagnosis of cancer. The osseous metastatic lesions do not need to be biopsied.
* Patients with multiple myeloma are eligible for the study.
* Patient has 1-3 major painful osseous metastases (target lesions) from any primary cancer or unknown primary cancer.
* Long bone target lesions must have a Mirels fracture score of ≤ 7.
* Patients with spinal cord compression from vertebral body metastases are not eligible.
* Target lesions have not previously been treated with radiation.
* Radiation oncologist determines that the patient is medically able to undergo palliative radiation therapy.
* Patient has target lesions that are radiographically consistent with metastatic disease on CT, MR, or PET CT obtained within 8 weeks of treatment.
* Persistent distinguishable pain associated with target sites to be treated.
* Patient average BPI pain score for last 72 hours at specified location is > 3 (0-10 scale)
* Patients may have additional non-painful or minimally painful osseous metastases (if patient has pain from additional sites, the pain from the additional sites must be evaluated as being less intense by at least 2 points on the BPI compared to the site(s) treated)
* The patient may have previously been treated with radiation therapy to other body sites, but not to the target lesions.
* The patient may have previously or currently be undergoing chemotherapy or bisphosphonate therapy.
* The patient will be able understand English (or a medical interpreter for their native language must be available for all study visits).
* 18 years of age or older.
* Life expectancy > 12 weeks.
* Able and willing to answer simple survey questionnaires.
* Able and willing to keep a logbook of analgesic use (with or without assistance).
* Willing to return to clinic for follow-up visits after first treatment.
* Signed study-specific informed consent form

Exclusion Criteria:

* Inability to lie flat on table for treatment
* Patient with < 12 weeks life expectancy
* Systemic radionuclide delivery within 30 days prior to treatment
* Epidural compression of spinal cord or cauda equine
* Spinal canal compromise > 25%
* Unstable spine requiring surgical stabilization
* Target lesions have previously been treated with radiation.
* Tumor located within 5mm of spinal cord or cauda equina.
* A serious uncontrolled medical disorder that, in the opinion of the Investigator, would impair the ability of the patient to receive protocol therapy.
* Pregnant and breastfeeding women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Read, MD, Study Chair — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 Patients were prospectively enrolled on a pilot clinical trial between 2011 and 2014. Patients were required to have biopsy-proven cancer with 1-3 painful osseous metastases, recent diagnostic imaging demonstrating metastatic disease, and persistent distinguishable pain at the target site(s) with an average pain score of 3 or greater
Groups:
- STAT RT Planning and Delivery Workflow: single arm
  STAT RT planning and delivery workflow: -Patients will receive simulation, planning, quality assurance, and their first treatment in a single day using the STAT RT workflow.
  * Patients will receive a total of 1-5 fractions of high dose palliative radiation therapy via TomoTherapy consisting of 5-10 Gray per fraction.
  * Data will be collected to evaluate the effectiveness of our novel image co-registration techniques, CT-detector-based exit dose calculations, and infrared patient position monitoring. These novel techniques for image co-registration, radiation dose calculations, and patient position monitoring will not alter or replace standard of care techniques.
Period: Overall Study
Arm/Group | STAT RT Planning and Delivery Workflow
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response, Partial Response, or Stable Pain After Receiving Treatment Via the STAT RT Workflow at 12-months
Description: The Brief Pain Inventory (BPI) and Oral Morphine Equivalent Doses (OMED) were used to categorize the number of participants who had a Complete Response (no pain), Partial Response (pain reduction), Stable Pain (no change in pain), and Pain Progression at 12 months after receiving treatment via the STAT RT workflow.
Time Frame: 12 months after treatment
Population: The Brief Pain Inventory (BPI) and Oral Morphine Equivalent Doses (OMED) were used to categorize the number of participants who had a Complete Response (no pain), Partial Response (pain reduction), or Stable Pain (no change in pain) at 12 months after receiving treatment via the STAT RT workflow.
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 9

2. Secondary Outcome: Number of Participants With Treatment Toxicity
Description: Toxicity will be assessed by CTCAE Version 4.0 Toxicity will be assessed up to 12 months after treatment.
Time Frame: 12 months after treatment
Population: Number of subjects with Grade 3 or higher adverse events within 12 months after initial treatment. No serious AEs reported; all AEs were grade 2 or less. Additional AE details found in published article.
Measure: Number; unit: participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
participants | 0

3. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 1 Week Post Treatment
Description: The patient's quality of life function will be assessed using the Brief Pain Inventory (BPI) 1 week post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 1 Week Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 19

4. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 4 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Brief Pain Inventory (BPI) 4 weeks post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 4 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 21

5. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 8 Weeks After Initial Treatment
Description: The patient's quality of life function will be assessed using the Brief Pain Inventory (BPI) 8 weeks post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 8 weeks post initial treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

6. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 12 Weeks Post Initial Treatment
Description: The patient's quality of life and function will be assessed using the Brief Pain Inventory (BPI) 12 weeks post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 12 weeks post treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

7. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 6 Months After Initial Treatment
Description: the patient's quality of life and function will be assessed using the Brief Pain Inventory (BPI) 6 months post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 6 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 13

8. Secondary Outcome: Number of Participants With an Improved Quality of Life Function Score at 12 Months After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Brief Pain Inventory (BPI) 12 months post treatment. Min-'0'/'Does not interfere'; Max-'10'/'Completely interferes.' ; Worst Pain Score: 1-4=Mild Pain, Worst Pain Score 5-6=Moderate Pain. Worst Pain Score 7-10=Severe Pain.
Time Frame: 12 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 10

9. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 1 Week Post Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 1 week post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 1 week post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 19

10. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 4 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 4 weeks post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 4 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 21

11. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 8 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 8 weeks post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 8 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

12. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 12 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 12 weeks post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

13. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 6 Months After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 6 months post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 6 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 13

14. Secondary Outcome: Patient Quality of Life and Function (FACT-BP) Assessed 12 Months After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-BP) survey 12 months post treatment. Min-'0'/'Not at all' and Maximum 4+ 'Very much.' Items scored per FACT_BP Scoring guidelines version 4; Score Range 0-60; The higher the score, the better QOL function.
Time Frame: 12 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 10

15. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 1 Week After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 1 week post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 1 week post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 19

16. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 4 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 4 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 4 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 21

17. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 8 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 8 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 8 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

18. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 12 Weeks After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 12 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 12 weeks post treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 15

19. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 6 Months After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 6 months post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 6 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 13

20. Secondary Outcome: Patient Quality of Life and Function (FACT-G) Assessed 12 Months After Initial Treatment
Description: The patient's quality of life and function will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) survey within 12 months post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; 28 questions total are broken into 4 categories scoring ranges 0-24 or 0-28 (depending on the category). Total score is ranged 0-108; Higher the score, the better quality of life (QOL).
Time Frame: 12 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 10

21. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 1 Week After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 1 week post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 1 week post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 19

22. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 4 Weeks After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 4 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 4 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 21

23. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 8 Weeks After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 8 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 8 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 14

24. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 12 Weeks After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 12 weeks post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 13

25. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 6 Months After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 6 months post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 6 months post treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 13

26. Secondary Outcome: Patient Quality of Life and Function (FACIT-TS-BTCSQ) Assessed 12 Months After Initial Treatment
Description: Estimate patient satisfaction with the STAT RT workflow using Functional Assessment of Chronic Illness Therapy-Bone Treatment Convenience and Satisfaction Questionnaire (FACIT-TS-BTCSQ). Satisfaction will be assessed within 12 months post treatment. Min-'0'/'Not at All'; Max-'4'/'Very Much'; FACIT-TS-BTCSQ Baseline Scoring Guidelines (Version 4) includes sub of individual items multiplied by 13 to give score; The higher the score, the higher the quality of life (QOL).
Time Frame: 12 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | STAT RT Planning and Delivery Workflow
Number analyzed (Participants) | 28
Participants | 9

ADVERSE EVENTS:
Time Frame: 30 days following last study treatment.
Description: Per protocol, treatment may continue for 2 to 5 fractions depending of the clinical situation. Most subjects will receive treatments for less than 1 week, however, all treatments must be completed within 21 days. AEs will be collected for 30 days following the last treatment.
Arm/Group | STAT RT Planning and Delivery Workflow
All-Cause Mortality (participants affected / at risk) | 14/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 12/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAT RT Planning and Delivery Workflow (N=28)
Fatigue (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-03-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT01391234/Prot_SAP_000.pdf
  • Informed Consent Form (2014-04-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT01391234/ICF_001.pdf